CLINICAL TRIAL: NCT00513045
Title: A Self-Help Method for Nightmares
Acronym: Nightmares
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht University (Other)
Collaborators: Fonds Psychische Gezondheid (Other)
Responsible Party: Utrecht University, Utrecht University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FPG20066126
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Nightmares
Keywords: Nightmares; treatment; self-help

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IRT (Experimental): Intervention based on Imagery Rehearsal Therapy
  Interventions: Behavioral: IRT
- Exposure (Active Comparator): Treatment based on exposure
  Interventions: Behavioral: Exposure
- Nightmare diary (No Intervention): Recording nightmares in a diary
- Waiting list (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: IRT — Cognitive behavior intervention
  Arms: IRT
Behavioral: Exposure — Exposure intervention
  Arms: Exposure

SUMMARY:
The objective of this study is to validate a newly designed self-help treatment for nightmares. This self-help treatment is based on Imagery Rehearsal Therapy. This treatment will be validated in comparison to an exposure treatment a diary condition and a waiting list condition.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from Nightmares
* Access to internet
* A valid e-mail address
* Be able to understand Dutch

Exclusion Criteria:

* Severe posttraumatic complaints
* Severe depression
* High anxiety ratings
* In therapy for post traumatic stress disorder
* Being suicidal
* Schizophrenic or having a psychosis episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Nightmare frequency | 1 year
Nightmare distress | 1 year

SECONDARY OUTCOMES:
Sleep quality | 1 year
Sleep complaints | 1 year
Anxiety ratings | 1 year
Posttraumatic complaints (low - moderate - high) | 1 year
Depression ratings | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van den Bout, Prof. dr., Study Director — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Related Info — http://www.nachtmerries.org